CLINICAL TRIAL: NCT05922709
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamic Profiles Following Single and Multiple Doses and Food Effect of CS12192 Capsules in Healthy Adult Chinese Subjects
Brief Title: A Clinical Trial of CS12192 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS12192-101
Record Dates: First submitted 2023-06-07; First posted 2023-06-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: healthy

STUDY DESIGN:
Intervention Model Description: The study consists of 3 parts: single ascending dose (SAD), multiple ascending dose (MAD) and food effect (FE). Both SAD and MAD study use a randomized, double-blind, placebo-controlled dose-escalation design. The FE study use a randomized, open-label, two-period, two-crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- CS12192 Cohort 1 (Experimental): Subjects receive a single dose of 50 mg CS12192 or matching placebo.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 2 (Experimental): Subjects receive a single dose of 150 mg CS12192 or matching placebo.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 3 (Experimental): Subjects receive a single dose of 200 mg CS12192 or matching placebo.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 4 (Experimental): Subjects receive a single dose of 300 mg CS12192 or matching placebo.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 5 (Experimental): Subjects receive a single dose of 400 mg CS12192 or matching placebo.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 6 (Experimental): Subjects receive 200 mg CS12192 or matching placebo for 7 days, twice daily (every 12 h) from Day 1 to Day 6, and once on Day 7.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 7 (Experimental): Subjects receive 300 mg CS12192 or matching placebo, twice daily (every 12 h) from Day 1 to Day 6, and once on Day 7.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 8 (Experimental): Subjects receive 400 mg CS12192 or matching placebo for 7 days, twice daily (every 12 h) from Day 1 to Day 6, and once on Day 7.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule
- CS12192 Cohort 9 (Experimental): Subjects receive a single dose 400 mg CS12192 in either the fasted or fed state for two periods.
  Interventions: Drug: CS12192 capsule
- CS12192 Cohort 10 (Experimental): Subjects receive a single dose of 600 mg CS12192 or matching placebo.
  Interventions: Drug: CS12192 capsule; Drug: Placebo capsule

INTERVENTIONS:
Drug: CS12192 capsule — Participants receive CS12192 orally single or multiple doses
Drug: Placebo capsule — Participants receive placebo matching CS12192 orally single or multiple doses
  Arms: CS12192 Cohort 1; CS12192 Cohort 10; CS12192 Cohort 2; CS12192 Cohort 3; CS12192 Cohort 4; CS12192 Cohort 5; CS12192 Cohort 6; CS12192 Cohort 7; CS12192 Cohort 8

SUMMARY:
The study is to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic profiles of CS12192 after single or multiple oral administration, as well as the food effect on the pharmacokinetics in healthy subjects.

DETAILED DESCRIPTION:
This study consists of 3 parts: single ascending dose (SAD), multiple ascending dose (MAD) and food effect (FE). Both SAD and MAD study are randomized, double-blind, placebo-controlled design. The FE study use a randomized, open-label, two-period, two-crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, both male and female.
* Between18 and 45 years of age (inclusive) at screening visit.
* BMI between 19.0-26.0 kg/m2 (including critical value) at screening visit and baseline visit, male subjects' body weight ≥ 50 kg, female subjects' body weight ≥45 kg.
* All subjects and female partners of male agree to use medically recognized effective contraceptive measures (including physical contraception, surgical contraception, abstinence, etc.) from the start of signing informed consent form to 3 months after the last dose.
* Subjects voluntarily participate in the study and sign informed consent form.

Exclusion Criteria:

* History of clinically significant drug allergy or atopic allergic diseases (asthma, urticaria, eczematous dermatitis) or drug allergy to investigational products or similar investigational products.
* History of cardiovascular system, endocrine system, nervous system disease or lung, hematological, immunological, psychiatric diseases and metabolic abnormalities.
* History or surgical history of gastrointestinal, hepatic, or renal disease that can affect drug absorption or metabolism within 6 months prior to the screening visit (except uncomplicated appendectomy and hernia repair).
* History of active tuberculosis, or positive tuberculosis screening at screening visit.
* History of any recurrent bacterial, fungal or viral infections (≥3 attacks in the past year, except the common cold), or active infections requiring treatment at screening visit, or history of infection requiring intravenous anti-infective drugs or hospitalization ≤8 weeks before randomization, or history of infection requiring oral anti-infective drugs ≤2 weeks before randomization.
* Uncured diarrhea before randomization, or history of diarrhea within 7 days before planning dosing.
* Use of any prescription drugs, over-the-counter drugs, any vitamin products or Chinese herbal medicines within 1 month before randomization.
* History of drug abuse.
* Inability to tolerate venipuncture, or history of fainting or halo.
* Participation in interventional clinical study (device or drug) within 3 months prior to randomization, or taking investigational product within 3 months prior to randomization , or remaining within 5 half-lives of drug, whichever is longer.
* Blood donation or significant blood loss (>300 mL) within 3 months prior to randomization.
* Pregnant or lactating females, or female subjects with serum pregnancy test human chorionic gonadotropin (HCG) ≥5 mIU/mL.
* History of regular alcohol consumption, drinking more than 7 cups per week for females or 14 cups per week for males (1 cup= 100 mL wine = 285 mL beer = 25 mL spirits) within 3 months before randomization; or taking any products containing alcohol within 48 hours before the first dose; or having a positive alcohol breath test before randomization.
* Smoking more than 5 cigarettes or equivalent per day within 3 months prior to randomization or inability to refrain from smoking during the trail.
* Excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups) per day within 14 days before randomization, or tea, coffee, caffeinated beverages or foods within 48 hours before randomization.
* Consumption of grapefruit or beverages or foods containing its ingredients within 14 days before randomization.
* Glomerular filtration rate (eGFR) <80 mL/min at screening visit and baseline visit (calculating by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation for serum creatinine, age, and sex).
* Abnormal results in medical history inquiry, vital signs, physical examination, chest X-ray, and clinical laboratory tests are clinically significant.
* QTcF≥450 ms or other clinically significant abnormality as judging by the investigator on 12-lead ECG at screening visit and baseline visit.
* Human immunodeficiency virus antibody (HIV) cannot provide negative reports at screening visit.
* Syphilis serology, hepatitis B virus surface antigen (HBsAg), hepatitis B virus-DNA quantification, or hepatitis C virus antibody (HCV-Ab) positive at screening visit.
* Positive urine drug screening (morphine, methamphetamine, ketamine, ecstasy, marijuana, cocaine) before randomization.
* Need or plan to engage in strenuous physical activity or exercise during the study.
* Inability to tolerate high-fat and high-fever meal (only for fed study).
* Subjects with dysphagia.
* Other conditions considered inappropriate for participation in the study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
the Number of Adverse Events (AEs) | up to 14 days
  To investigate the safety and tolerability by assesment of AEs following administration.
Pharmacokinetic parameters - Area Under the Curve(AUC) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses. From time 0 to 48 hours after the last dose for food effect study.
  Area Under the Plasma Concentration-time Curve of CS12192.
Pharmacokinetic parameters - Peak Plasma Concentration (Cmax) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses. From time 0 to 48 hours after the last dose for food effect study.
  Maximum Observed Plasma Concentration of CS12192.
Pharmacokinetic parameters - Time of peak concentration(Tmax) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses.From time 0 to 48 hours after the last dose for food effect study. From time 0 to 48 hours after the last dose for food effect study.
  Time to reach maximum observed plasma concentration of CS12192.
Pharmacokinetic parameters - Plasma Elimination Half-Life(t1/2) | From time 0 to 48 hours for single dose. From time 0 to 48 hours after the last dose for multiple doses.From time 0 to 48 hours after the last dose for food effect study. From time 0 to 48 hours after the last dose for food effect study.
  Plasma Elimination Half-Life of CS12192.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No